CLINICAL TRIAL: NCT00248807
Title: Systemic Hemodynamics and Cerebral Blood Flow in Persons With Tetraplegia
Brief Title: A Study of Blood Pressure and Blood Supply to the Brain in Persons With a Spinal Cord Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B3346-V; 00517 (Other: JJP VAMC IRB)
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Orthostatic Hypotension; Spinal Cord Injuries
Keywords: Blood Pressure, Low; Hypotension, Postural; Injuries, Spinal Cord; Spinal Cord Transection; Spinal Cord Trauma
MeSH Terms: conditions — Hypotension, Orthostatic; Spinal Cord Injuries; Hypotension

ARMS (4):
- ARM 1 (Placebo Comparator): Head-up tilt maneuver without drug in subjects with spinal cord injury
  Interventions: Other: Head up tilt (HUT)
- ARM 3 (Placebo Comparator): Head-up tilt maneuver without drug in able-bodied controls
  Interventions: Other: Head up tilt (HUT)
- ARM 2 (Active Comparator): Head-up tilt maneuver with an angiotensin converting enzyme inhibitor (1.25 mg enalaprilat) in subjects with spinal cord injury
  Interventions: Drug: 1.25 mg enalaprilat IV; Other: Head up tilt (HUT)
- ARM 4 (Active Comparator): Head-up tilt maneuver with an angiotensin converting enzyme inhibitor (1.25 mg enalaprilat) in able-bodied controls.
  Interventions: Drug: 1.25 mg enalaprilat IV; Other: Head up tilt (HUT)

INTERVENTIONS:
Drug: 1.25 mg enalaprilat IV — an angiotensin converting enzyme (ACE) inhibitor given to lower blood pressure (BP) and measure cerebral blood flow (CBF)
  Arms: ARM 2; ARM 4
Other: Head up tilt (HUT) — 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow.

SUMMARY:
The purpose of this study is to determine how blood pressure and blood flow are controlled during head-up tilt in a semi-upright position. In this investigation we are studying blood pressure and blood flow to the brain, with and without a medication which lowers blood pressure (Vasotec). We will determine how persons with a spinal cord injury are able to maintain blood flow to the brain (not get dizzy) as they assume a more upright position and their blood pressure decreases.

DETAILED DESCRIPTION:
Individuals with tetraplegia lack normal sympathetic nervous system regulation of blood pressure and, therefore, relative hypotension is a common occurrence. This hypotension may be more pronounced with postural stress. Loss in mental acuity and sometimes even consciousness is an associated symptom of postural hypotension in individuals with tetraplegia.

There is some evidence to suggest that although mean arterial blood pressure (MAP) is relatively low in these individuals, middle cerebral arterial blood flow (CBF) may be maintained. Consequently, individuals with chronic tetraplegia often compensate and are stable in the seated upright position.

Autoregulation of CBF has been defined as the stability of cerebral blood flow throughout a range of systemic blood pressures (MAP). This proposal will examine systemic hemodynamics and middle cerebral artery blood flow during HUT with and without Vasotec, an angiotensin II inhibitor. By partially or completely ablating the renin-angiotensin system, which is postulated to play a major role in blood pressure regulation, the potential dissociation between systemic blood pressure and middle cerebral artery blood flow, in individuals with tetraplegia, may be demonstrated. The aim is to determine whether persons with chronic tetraplegia are able to maintain similar CBF, or similar CBF changes, as able-bodied controls despite a greater decrease in MAP to the same hypotensive challenge. The relationship between MAP and CBF has not been defined in this population. Understanding this relationship may lead to improved screening and treatment for prevention of postural hypotension in persons with tetraplegia.

ELIGIBILITY:
Inclusion Criteria:

* Duration of spinal cord injury (SCI) at least 1 year
* Level of SCI C4-8 and T6 and below
* matched non-SCI subjects
* Chronological age between 18-65 years
* Euhydration: Subjects will be instructed to avoid caffeine and alcohol and to maintain normal salt and water intake for several days prior to study.

Exclusion Criteria:

* Known heart and/or blood vessel disease
* Dehydration
* High blood pressure
* Kidney disease
* Diabetes mellitus
* Prescribed ACE inhibitors
* Acute Infection
* Smoking
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2009-05 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Wecht, EdD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- [Result] Handrakis JP, DeMeersman RE, Rosado-Rivera D, LaFountaine MF, Spungen AM, Bauman WA, Wecht JM. Effect of hypotensive challenge on systemic hemodynamics and cerebral blood flow in persons with tetraplegia. Clin Auton Res. 2009 Feb;19(1):39-45. doi: 10.1007/s10286-008-0496-6. Epub 2008 Oct 11. PMID 18850311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment has been completed.
Pre-assignment Details: All subjects recruited completed all testing procedures.
Groups:
- Subjects With Spinal Cord Injury (SCI): Subjects with SCI underwent a 45 degree head-up tilt maneuver to lower blood pressure and measure cerebral blood flow with and without enalaprilat (1.25 mg).
- Subjects Without SCI (Non-SCI): Subjects without SCI (non-SCI) underwent a 45 degree head-up tilt maneuver to lower blood pressure and measure cerebral blood flow with and without enalaprilat (1.25 mg).
Period: Overall Study
Arm/Group | Subjects With Spinal Cord Injury (SCI) | Subjects Without SCI (Non-SCI)
Started | 19 | 11
Completed | 19 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects With Spinal Cord Injury: Subjects with spinal cord injury underwent a 45 degree head-up tilt maneuver to lower blood pressure and monitor cerebral blood flow on 2 study visits. The first visit subject underwent the head-up tilt maneuver without drug and on the second visits subject underwent the head-up tilt maneuver following oral administration of an angiotensin converting enzyme inhibitor (ACE: 1.25 mg enalaprilat).
- Non-spinal Cord Injured Subjects: Non-spinal cord injured subjects underwent a 45 degree head-up tilt maneuver to lower blood pressure and monitor cerebral blood flow on 2 study visits. The first visit subject underwent the head-up tilt maneuver without drug and on the second visits subject underwent the head-up tilt maneuver following oral administration of an angiotensin converting enzyme inhibitor (ACE: 1.25 mg enalaprilat).
- Total: Total of all reporting groups
Arm/Group | Subjects With Spinal Cord Injury | Non-spinal Cord Injured Subjects | Total
Number analyzed (Participants) | 19 | 11 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 11 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11) | 35 (12) | 39 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 16 | 9 | 25
Region of Enrollment [Number; unit: participants]
  United States | 19 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure during head-up tilt in subjects with spinal cord injury without drug intervention
Time Frame: acute testing
Population: convenience sample
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- ARM 1: 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow in subjects with spinal cord injury without drug
- ARM 2: 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow in able-bodied control subjects without drug
- ARM 3: 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow in subjects with spinal cord injury following intravenous administration of an angiotensin converting enzyme inhibitor (1.25 mg enalaprilat).
- ARM 4: 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow in able-bodied control subjects following intravenous administration of an angiotensin converting enzyme inhibitor (1.25 mg enalaprilat).
Arm/Group | ARM 1 | ARM 2 | ARM 3 | ARM 4
Number analyzed (Participants) | 19 | 11 | 19 | 11
mmHg | 123 (37) | 125 (15) | 119 (26) | 122 (14)

2. Secondary Outcome: Cerebral Blood Flow
Description: Measurement of middle cerebral artery blood flow velocity supine and during head-up tilt
Time Frame: acute testing
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | ARM 1 | ARM 2 | ARM 3 | ARM 4
Number analyzed (Participants) | 19 | 11 | 19 | 11
cm/sec | 45.95 (8.71) | 42.52 (15.69) | 46.93 (7.66) | 37.38 (4.44)

ADVERSE EVENTS:
Groups:
- ARM 1: 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow in subjects with spinal cord injury.
- ARM 2: 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow in able-bodied controls.
- ARM 3: 1.25 mg enalaprilat IV and 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow in subjects with spinal cord injury.
- ARM 4: 1.25 mg enalaprilat IV and 45 degree head-up tilt to lower blood pressure and measure cerebral blood flow in able-bodied controls.
Arm/Group | ARM 1 | ARM 2 | ARM 3 | ARM 4
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/19 | 0/11
Other Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/19 | 0/11

LIMITATIONS AND CAVEATS:
Did not assess carbon dioxide levels or the severity of spinal cord injury, which may have contributed to the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No